CLINICAL TRIAL: NCT03227575
Title: Effects of Brisk Walking and Regular Intensity Exercise Interventions on Glycemic Control
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Original PI changed institutions and COVID
Sponsor: Plymouth State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0001
Record Dates: First submitted 2017-06-28; First posted 2017-07-24 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Metabolic Syndrome; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Post-Meal Walking Group (Experimental): Following a 30-minute digestion period, the Post-Meal Walking Group will be instructed to walk following breakfast, lunch, and dinner at least 4 times per week (180 minutes of moderate intensity exercise/week). Participants will walk at a brisk pace for 15 minutes, as demonstrated in a previous study. A Garmin VivoFit activity monitor will measure their physical activity across the four-week intervention. The Garmin VivoFit activity monitor must be returned during the "Follow-up Study Visit".
  Interventions: Behavioral: Exercise Intervention
- Traditional Exercise Group (Experimental): The Traditional Exercise Group will perform aerobic and light resistance training exercise over the 4-week intervention. A group of trained Exercise and Sports Physiology students will conduct the aerobic exercise and light resistance training program three times per week (180 minutes of moderate to high intensity exercise/week). Garmin VivoFit activity monitors will measure their physical activity across the four-week intervention. The Garmin VivoFit activity monitor must be returned during the "Follow-up Study Visit".
  Interventions: Behavioral: Exercise Intervention
- Case Control Group (No Intervention): The participant will be instructed to maintain their current diet and levels of physical activity for four weeks. Participants in this group will wear an ambulatory blood pressure monitor at baseline and at follow-up. Any change in diet and physical activity level might significantly affect the study results. The Control Group will maintain their current lifestyle for four weeks. Garmin VivoFit activity monitors will measure their physical activity throughout the 4-week intervention. The Garmin VivoFit activity monitor must be returned during the "Follow-up Study Visit".

INTERVENTIONS:
Behavioral: Exercise Intervention — The use of exercise to improve glycemic responses in young adults who are at risk for Metabolic Syndrome.
  Arms: Post-Meal Walking Group; Traditional Exercise Group

SUMMARY:
Physical activity is shown to positively reduce the risk of developing both cardiovascular disease and type 2 diabetes. Current guidelines recommend 30-60 minutes of moderate intensity cardiorespiratory exercise five days per week. However, studies report that <40% of young adults 18-24 years achieve the recommended weekly physical activity guidelines, and close to 40% of young adults are overweight or obese. Traditional aerobic exercise and high intensity exercise have been shown to improve glycemic control in young and middle-aged sedentary adults, however, long term implementation of such exercise regimens are difficult. Recent evidence suggests that short bouts (15 minutes) of moderate intensity walking following a meal, significantly improves glycemic control in older adults with impaired glucose control. Due to the low burden of walking on participants, moderate intensity post-meal walking might be a better alternative exercise intervention to improve overall health in a sedentary population. Therefore, the purpose of this pilot proposal is to determine if 15 minutes of post-meal walking is an effective intervention to improve glycemic control in sedentary young adults at risk for developing MetS. Additionally, the study will investigate whether ambulatory blood pressure profiles in obese young adults are disrupted.

DETAILED DESCRIPTION:
Sedentary young adults (18-39 years) will be recruited from the community and surrounding areas of Plymouth, NH. In order to be included in the study sample, participants must meet the following criteria: a BMI > 26.9, body fat % >19.9% for men, body fat greater than 31.9 for women, and who do not participate in regular physical activity. Participants will be free of any known signs and symptoms of cardiovascular disease, diabetes, chronic kidney disease, and cancer.

Questionnaires The investigators will utilize two questionnaires for the study. Investigators will use a Health History Questionnaire to assess baseline health information. Investigators will also use the International Physical Activity Questionnaire to assess current physical activity status.

Waist Circumference, Height, Body Composition, and Weight Investigators will measure waist circumference using a Gulick measuring tape. Investigators will collect height using Stadiometer scale. Weight and body composition will be collected using a Tanita Scale, which assesses weight and body composition

Blood Pressure Blood pressure will be measured utilizing manometry (blood pressure cuff), which is traditionally used by clinicians to measure blood pressure.

Garmin VivoFit Activity Monitor A Garmin VivoFit activity monitor will be used to collect daily exercise, track steps per day, and heart rate. The monitor is worn on the wrist and allows for the accurate measurement of daily physical activity, steps per day, and daily heart rate. These variables and other measurement variables from daily activity, heart rate, and daily steps will be tracked with the watch.

IV Catheter Placement An intravenous (IV) catheter will be placed into a superficial vein either at the elbow (normally where blood is drawn) or vein near the wrist (secondary option for venous blood sampling). Catheter placement will be performed by Dr. Michael Brian, who has been previously trained in phlebotomy and proper IV catheter insertion at the University of Delaware. The IV catheter is vital for completing successive blood draws during the testing visit. Professor Sandra Gamble, of the Nursing Department, will assist during data collections to ensure safe blood collections.

75g Glucose Drink A standardized 75g glucose drink will be utilized to as part of the oral glucose tolerance tests, which is a test to assess the body's response to glucose.

Blood Sample Processing A OneTouch portable blood glucose monitor will be used to assess blood glucose from whole blood samples during the study visit. The remaining whole blood will be centrifuged and the extracted serum will be stored for future insulin analysis. All serum samples will be stored in a -80 freezer until analysis.

24-hour Blood Pressure Monitoring The investigators will utilize a 24-hour blood pressure monitor (Oscar 2-SunTech Blood Pressure Monitor, Morrisville, NC, USA) to measure blood pressure over a 24-hour period. The cuff will be fitted to the participant's arm and will take blood pressure every 20 minutes during the daytime and every 30 minutes during the night time. Throughout the 24-hour period, participants will be asked to maintain their normal daily routines.

Questionnaires (Appendix B) We will utilize two questionnaires for the study. We will use a Health History Questionnaire to assess baseline health information. We will also use the International Physical Activity Questionnaire to assess current physical activity status.

Waist Circumference, Height, Body Composition, and Weight We will measure waist circumference using a Gulick measuring tape. We will collect height using Stadiometer scale. Weight and body composition will be collected using a Tanita Scale, which assesses weight and body composition.

24-hour Blood Pressure Monitoring We will utilize a 24-hour blood pressure monitor (Oscar 2-SunTech Blood Pressure Monitor, Morrisville, NC, USA) to measure blood pressure over a 24-hour period. The cuff will be fitted to the participant's arm and will take blood pressure every 20 minutes during the daytime and every 30 minutes during the night time. Throughout the 24-hour period, participants will be asked to maintain their normal daily routines.

Garmin VivoFit Activity Monitor A Garmin VivoFit activity monitor will be used to collect daily exercise, track steps per day, and heart rate. The monitor is worn on the wrist and allows for the accurate measurement of daily physical activity, steps per day, and daily heart rate. These variables and other measurement variables from daily activity, heart rate, and daily steps will be tracked with the watch.

IV Catheter Placement An intravenous (IV) catheter will be placed into a superficial vein either at the elbow (normally where blood is drawn) or vein near the wrist (secondary option for venous blood sampling). Catheter placement will be performed by Dr. Michael Brian, who has been previously trained in phlebotomy and proper IV catheter insertion at the University of Delaware. The IV catheter is vital for completing successive blood draws during the testing visit.

75g Glucose Drink A standardized 75g glucose drink will be utilized to as part of the oral glucose tolerance tests, which is a test to assess the body's response to glucose.

Blood Sample Processing Whole blood will be spun down to separate serum and red blood cells. The serum will be extracted and stored for future insulin analysis. All serum samples will be stored in a -80 freezer until analysis.

Insulin Analysis In collaboration with Dr. Heather Doherty, insulin analysis will be performed on stored serum blood samples using a Human Insulin ELISA kit. Dr. Doherty has offered to assist and guide Dr. Brian in the proper analysis insulin levels measured from our study population. The analysis will be completed following the completion of the study.

24-hour Continuous Glucose Monitor (CGM) A subcutaneous (just below the skin) Dexcom G5 Sensor (Dexcom; San Diego, California) will be placed on the abdomen by Dr. Michael Brian. The sensor measures glucose levels in the body every 5 minutes over a 24-hour period for 7 days. Participants will be trained how use the equipment, which requires a participant to calibrate the sensor two times daily by measuring their blood glucose through a finger prick.

Protocol All participants will complete an informed consent, and then screened prior to being enrolled into the study. As part of the initial screening visit, participants will complete a health history questionnaire, International Physical Activity Questionnaire (to assess current sedentary status), waist circumference measurement, height & weight measures, body composition, and resting blood pressure. Participants will then be randomized into two study groups (Post-Meal Walking Group, Traditional Exercise Group).

Continuous Glucose Monitoring Visit

Prior to the "Baseline Study Visit," participants will come to the Exercise and Sports Physiology Research Laboratory (Draper & Maynard Building, room 417) for CGM training and subcutaneous sensor insertion. Participants will receive training on proper care of the CGM unit, calibration techniques, and proper lancet disposal in a Sharps container. Following CGM sensor insertion and training, participants will be allowed to leave for 1.5 hours while the sensor warm-ups and then return to the laboratory for sensor calibration. After sensor calibration, participants will wear the CGM unit for the next 6 days. The total visit will take approximately 2.5 hours (including the warm-up period).

Baseline Study Visit

Six days after the CGM insertion, participants will arrive 8 hours fasted to the Exercise and Sports Physiology Research Laboratory (D&M 417) on the morning of the study visit. Participants will be asked to complete a three-day diet record. Baseline measurements of height, weight, waist circumference, blood pressure, heart rate, and body composition will be made. Following the baseline measurements, Michael Brian (PhD) will insert a catheter into the arm of the participant, leaving a small flexible tubing in the arm to collect blood samples throughout the protocol. A baseline blood collection will be performed to assess fasting insulin levels in the body.

Participants will then complete an oral glucose tolerance test. Participants will consume a 75g glucose drink to measure the participant's glycemic response. The glucose drink simulates an individual consuming a high sugar load, like a soda. Blood samples will be collected at 30, 60, and 120-minute time points following glucose consumption. Following the completion of the oral glucose tolerance test, the catheter and CGM will be removed and vitals checked (blood pressure & heart rate). Participants will then be provided with a 24-hour blood pressure monitor to wear. The participants will return the blood pressure monitor the following day.

4-Week Exercise Intervention

Following the "Initial Study Visit," participants will be provided with detailed instructions for their intervention. Participants will be randomly divided into two groups: Post-Meal Walking Group and Traditional Exercise Control Group.

Throughout the 4-weeks, participants will be asked to continue their regular diet and daily levels of physical activity. They will be instructed that changing their diet or physical activity levels outside of the study can significantly impact the study results.

Post-Meal Walking Group

Following a 30-minute digestion period, the Post-Meal Walking Group will be instructed to walk following breakfast, lunch, and dinner at least 4 times per week (180 minutes of moderate intensity exercise/week). Participants will walk at a brisk pace for 15 minutes, as demonstrated in a previous study (5). A Garmin VivoFit activity monitor will measure their physical activity across the four-week intervention. The Garmin VivoFit activity monitor must be returned during the "Follow-up Study Visit".

Traditional Exercise Group

The Traditional Exercise Group will perform aerobic and light resistance training exercise over the 4-week intervention. A group of trained Exercise and Sports Physiology students will conduct the aerobic exercise and light resistance training program three times per week (180 minutes of moderate to high intensity exercise/week). Garmin VivoFit activity monitors will measure their physical activity across the four-week intervention. The Garmin VivoFit activity monitor must be returned during the "Follow-up Study Visit".

A general exercise prescription will be used to standardized all Traditional Exercise sessions.

Follow-up Study Visit

Participants will complete all of the measurements performed during the "Initial Study Visit" and all activity monitors will be collected.

Case Control Study

A case control study will be used to measure ambulatory 24-hour blood pressure monitoring in healthy sedentary controls. This will help in our attempt to determine whether 24-hour blood pressure control is disrupted in sedentary obese individuals.

After an initial screening visit, participants will wear an ambulatory blood pressure monitor for 24 hours, and return it the next day. The participants will be instructed to maintain their current diet and levels of physical activity for four weeks. Any change in diet and physical activity level might affect the study results. A Garmin VivoFit activity monitor will be provided to measure their physical activity over four weeks. At the end of the 4-week period, participants will have their 24-hour blood pressure measured again. The Garmin VivoFit activity monitor and 24-hour blood pressure cuff must be returned the day after the 24-hour blood pressure monitoring period.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 30
* Currently not physically active
* Free of any signs and symptoms of cardiovascular disease, diabetes, chronic kidney disease, and cancer.

Exclusion Criteria:

* Planning to become pregnant
* Any known signs and symptoms of cardiovascular disease, diabetes, chronic kidney disease, and cancer.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Determine whether ambulatory blood glucose control responses are improved following 28 days of exercise training (Post Training). | An average of 32 days will separate these two measurements.
  Examine blood glucose (mg/dL) responses during two oral glucose tolerance test (70g glucose drink). The first test will be measured at baseline (Base) and the second test will be measured following 28 days of exercise training. These two tests (Base vs Post Training) will be separated by an average of 32 days.
Determine whether serum insulin (IU/mL) responses are improved following 28 days of exercise training (Post Training). | An average of 32 days will separate these two measurements.
  Examine serum insulin (IU/mL) responses during two oral glucose tolerance tests (70g glucose drink). The first test will be measured at baseline (Base) and the second test will be measured following 28 days of exercise training. These two tests (Base vs Post Training) will be separated by an average of 32 days.

SECONDARY OUTCOMES:
Determine whether ambulatory blood pressure profiles are different following an average of 28 day exercise intervention compared to sedentary healthy controls. | An average of 28 days will separate these two measurements.
  We will exam ambulatory 24-hour blood pressure profiles in healthy sedentary young adults at baseline, and then re-measure ambulatory 24-hour blood pressure profiles during a follow-up visit. These will be compared to our obese young adults.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Draper & Maynard, Plymouth, New Hampshire
  - Plymouth State University, Plymouth, New Hampshire

IPD SHARING:
Plan to Share IPD: No